CLINICAL TRIAL: NCT03022318
Title: Short Term Effects of Carbidopa-levodopa in Neovascular AMD
Brief Title: Carbidopa-levodopa in Neovascular AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Snyder, Robert W., M.D., Ph.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-07

CONDITIONS: Age-related Macular Degeneration
Keywords: GPR143; PEDF; VEGF; LDOPA
MeSH Terms: conditions — Macular Degeneration | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- once daily (Experimental): carbidopa-levodopa 25-100 mg tablets once daily hs for up to 32 days
  Interventions: Drug: carbidopa-levodopa 25-100 mg tablets
- 3 times daily (Experimental): carbidopa-levodopa 25-100 mg tablets 3 times daily,in the morning, with supper and hs for up to 32 days
  Interventions: Drug: carbidopa-levodopa 25-100 mg tablets

INTERVENTIONS:
Drug: carbidopa-levodopa 25-100 mg tablets — See arm/group descriptions
  Other Names: Sinemet

SUMMARY:
From 3 large patient databases, patients diagnosed with AMD who have never taken levodopa(L-DOPA) containing medications have a mean age of diagnosis at 71 years. Patients who have been treated with L-DOPA containing medications have a mean age of diagnosis of AMD at 79 years.

L-DOPA binds to GPR143 in the retinal pigment epithelium, and releases PEDF, which protects the retina and downregulates VEGF, which is the cause of neovascularization.

The Investigators will evaluate the safety and tolerability of carbidopa-levodopa in patients with Neovascular AMD, and measure the effects on visual acuity and retinal abnormalities due to "wet" (neovascular) AMD.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the most common cause of blindness, in individuals over the age of 50, in the developed world. AMD becomes more common as people age and is more common in lightly pigmented individuals. AMD appears more common in patients with Parkinson's Disease than in those without. The AREDS nutritional supplements are effective in slowing the progress of intermediate AMD(5). Most AMD is "dry AMD", which progresses relatively slowly and may impair vision, but usually does not lead to legal blindness. There are two forms of AMD, "wet AMD" and geographic atrophy (GA), that can cause more profound vision loss. In aggregate, they occur in about 25% of patients with AMD. Wet AMD is due to new growth of abnormal blood vessels under the retina. The new blood vessels are believed to be due to an excessive release of vascular endothelial growth factor (VEGF) by the retinal pigment epithelium(RPE) cells. Wet AMD is now effectively treated with intraocular injections of VEGF inhibitors. Geographic Atrophy, the other form of advanced AMD, represents focal death of the RPE cells and overlying neurosensory retina. There is no current treatment for GA. It is suspected that GA is due in part to a localized inflammatory response, damage to RPE cells, and loss of RPE cell function. It may also be speculated that stimulation of RPE cells to release a potent neurotrophic factor, pigment epithelium derived factor (PEDF) may slow the progression of GA.

In 2008, Dr. Brian McKay identified a receptor, G protein coupled receptor #143(GPR143), on the surface of RPE cells and discovered that L-DOPA was the natural ligand or stimulator of GPR143. Dr McKay showed that treatment of RPE cells with exogenous L-DOPA resulted in the release of additional PEDF. In subsequent work, Dr. McKay's group also showed that L-DOPA stimulation of PEDF in RPE cells was also associated with a decrease in VEGF. Thus, Dr McKay hypothesized that exogenous L-DOPA may prevent the onset of AMD or progression to wet AMD.

In 2015, Dr McKay and his associates published a paper that showed that patients, who had been treated with L-DOPA, had a delay in the onset of AMD by 8 years, compared to patients who had not been treated with L-DOPA. In addition, those who had AMD and went on to develop wet AMD did so 5 years later than those with no history of L-DOPA treatment. L-DOPA is an intermediate in the pigmentation pathway. Dr McKay and his associates suggested that the reason darkly pigmented races do not get AMD nearly as frequently as lighter pigmented races is that they produce more pigment, and thus more L-DOPA to stimulate GPR143 on RPE cells. According to this hypothesis, the stimulated RPE cells release PEDF and decrease VEGF, which together are responsible for the protective effect.

Since there are no established animal models for AMD, and L-DOPA has a good safety profile in healthy volunteers and patients with Parkinson's disease, the Investigators propose a prospective experiment to determine the safety and tolerability of L-DOPA, in a population of patients with AMD. The participants will be made aware of potential side effects of L-DOPA, which are listed in the Informed Consent, during the consent process. Adverse events will be elicited by questioning the participants at each visit. The participants will also be advised to call the site if they have any medical problems between visits.

The Investigators will also use this study to examine whether L-DOPA has a positive effect on visual acuity and pathologic retinal changes of "wet" AMD. The parameters to be evaluated are best corrected ETDRS visual acuity, macular thickness by spectral domain optical coherence tomography (SD OCT), new blood (hemorrhage) by direct retinal examination, or subjective decrease in vision.

Pharmacology of L-DOPA and carbidopa:

L-DOPA is formed by 3-hydroxylation of tyrosine by tyrosine-3-monooxygenase (tyrosinase).(18) The primary metabolic pathway of L-DOPA is decarboxylation by amino acid decarboxylase to dopamine, which is responsible for most, but not all, of its pharmacologic effects and toxicity. When carbidopa is administered with L-DOPA, systemic levels of L-DOPA double and central nervous system (CNS) L-DOPA increases from about 1% of the administered dose to about 4%. Levodopa freely passes from the systemic circulation into the retina and brain, but dopamine and carbidopa do not. Adverse events are markedly decreased when carbidopa is administered with L-DOPA, because systemic levels of the toxic metabolite of L-DOPA, dopamine, are markedly reduced. In most patients, 25 mg of carbidopa is sufficient to control side effects of 100 mg of L-DOPA, primarily nausea, by 90%.

L-DOPA is the natural ligand for GPR143 in the RPE cells. The Investigators' intent is to increase the L-DOPA available to RPE surface receptors (GPR 143) while minimizing peripheral toxicity. This concept is unique, because all other uses of L-DOPA rely on CNS conversion of L-DOPA to dopamine, in order to produce the desired effect.

Excess VEGF is the mediator of the retinal neovascularization and other retinal pathological changes in "wet" AMD. Intraocular injections of anti-VEGF antibodies is the standard of care in "Wet" AMD. Several publications, including Lim et al, show that with careful monitoring of the visual acuity and retinas of patients with wet AMD, if there is no progression, there are no long-term adverse consequences of delaying initiation of anti-VEGF therapy for up to 4 weeks. The patients will be monitored at weekly intervals, for up to 4 weeks, for indications for initiation of anti-VEGF injections.

Criteria for anti-VEGF injections

This will be based on: weekly evaluation of ETDRS visual acuity (decrease of 5 letters from previous visit); increased macular thickness (compared to normal and previous visit as measured by OCT; new blood (hemorrhage) on direct retinal examination; or subjective decrease in vision. If any of these criteria are met, or if, in the opinion of the Ophthalmologist, the patient requires anti-VEGF therapy, the patient will have an anti-VEGF intraocular injection. If none of these criteria are met at visits 2, 3, or 4, with the patient agreement, anti-VEGF injection will not be done, and the patient will be reevaluated in 1 week. The patients will receive an anti-VEGF injection at the end of the 4th week if they have not received one earlier. Whenever a patient receives the first anti-VEGF injection, participation in this protocol will end. At that point, the patient will be able to enroll in Study 0002, Proof of Concept and Dose Ranging Study of carbidopa-levodopa in Neovascular AMD.

Treatments:

Randomized assignment to carbidopa-levodopa 25-100 mg tablets dosed hs or carbidopa-levodopa 25-100 mg tablets dosed 3 times daily, in the morning, with supper and hs. The second dosing regimen is the equivalent of a moderate dose of carbidopa-levodopa in patients with Parkinson's disease (maximum daily dose of levodopa 200-800 mg).

Number of participants: Up to 52 completed, randomized using a table of random numbers.

Informed Consent will be completed at the first visit. Duration: up to 32 days of treatment. Visits will occur at 5-8 day intervals. Overall trial duration for enrollment and treatment, screening 5 patients per week, will be approximately 10 months.

Primary Endpoint: A statistically significant improvement (5 letters) by carbidopa-levodopa treatment in ETDRS visual acuity.

Measurements:

Demographics at Visit 1; Medical History and Physical Examination at Visit 1; Electrocardiogram(ECG), complete blood count(CBC), Chem 20 and HbA1C at Visit 1; Vital signs at Visits 1,2,3,4 and 5; Non-directed assessment of adverse events at Visits 1,2,3,4 and 5. SD OCT at Visits 1,2,3,4,5; Pill count at Visits 2,3,4 and 5;

Statistics: Analysis of Variance with Independent Variables for each arm and comparing arms:

ETDRS visual acuity, central retinal (macular) thickness, presence of hemorrhage and duration of treatment prior to initiation of anti-VEGF (Vascular endothelial growth factor) intraocular injections.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of AMD with choroidal neovascularization (CNV) in one eye;
2. Not previously treated with anti-VEGF injections;
3. Normal or dry AMD of any grade in the second eye;
4. Age 50-85 years;
5. Willingness to maintain AREDS vitamin supplements throughout the study, or remain off these supplements for the duration of the study, if not taking them prior to the study;
6. Signed Informed Consent.

   -

Exclusion Criteria:

1. Any current use of L-DOPA containing medication or dopamine agonist medication, or any planned use of any of these agents, except for study medication, during the study;
2. Concurrent use of monoamine oxidase (MAO) inhibitors;
3. Any eye condition, disease, or history of trauma in either eye, which can impair vision, except cataract or cataract surgery;
4. Best Corrected Visual Acuity (BCVA )worse than 20/160 in the better eye;
5. Wet AMD in the second eye;
6. Neurologic conditions which can impair vision;
7. Parkinson's Disease;
8. Significant orthostatic hypotension, defined as a drop in systolic blood pressure, immediately upon changing from the supine to standing position, of >19 mmHg, or a symptomatic drop in systolic blood pressure, immediately upon changing from the supine to standing position;
9. Significant ECG abnormalities, as judged by the Investigator;
10. Estimated glomerular filtration rate (eGFR) <20 ml/min;
11. Liver enzymes >3 X the upper limit of normal;
12. HbA1C >9.0;
13. Any other significant lab abnormalities, as judged by the Investigator;
14. Women of childbearing potential;
15. Known retinal hemorrhage;
16. Subjects who are not fluent in English.

    -

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Snyder, MD, PhD, Principal Investigator — Robert W Snyder, MD, PhD, PC; Timothy C Fagan, MD, Study Director — Robert W Snyder, MD, PhD, PC
Locations (1):
- Robert W Snyder, MD, PhD, PC, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Jager RD, Mieler WF, Miller JW. Age-related macular degeneration. N Engl J Med. 2008 Jun 12;358(24):2606-17. doi: 10.1056/NEJMra0801537. No abstract available. PMID 18550876
- [Background] Bressler SB, Munoz B, Solomon SD, West SK; Salisbury Eye Evaluation (SEE) Study Team. Racial differences in the prevalence of age-related macular degeneration: the Salisbury Eye Evaluation (SEE) Project. Arch Ophthalmol. 2008 Feb;126(2):241-5. doi: 10.1001/archophthalmol.2007.53. PMID 18268216
- [Background] Ferrara N. Vascular endothelial growth factor and age-related macular degeneration: from basic science to therapy. Nat Med. 2010 Oct;16(10):1107-11. doi: 10.1038/nm1010-1107. No abstract available. PMID 20930754
- [Background] Lopez VM, Decatur CL, Stamer WD, Lynch RM, McKay BS. L-DOPA is an endogenous ligand for OA1. PLoS Biol. 2008 Sep 30;6(9):e236. doi: 10.1371/journal.pbio.0060236. PMID 18828673
- [Background] Falk T, Congrove NR, Zhang S, McCourt AD, Sherman SJ, McKay BS. PEDF and VEGF-A output from human retinal pigment epithelial cells grown on novel microcarriers. J Biomed Biotechnol. 2012;2012:278932. doi: 10.1155/2012/278932. Epub 2012 Apr 2. PMID 22547925
- [Background] Brilliant MH, Vaziri K, Connor TB Jr, Schwartz SG, Carroll JJ, McCarty CA, Schrodi SJ, Hebbring SJ, Kishor KS, Flynn HW Jr, Moshfeghi AA, Moshfeghi DM, Fini ME, McKay BS. Mining Retrospective Data for Virtual Prospective Drug Repurposing: L-DOPA and Age-related Macular Degeneration. Am J Med. 2016 Mar;129(3):292-8. doi: 10.1016/j.amjmed.2015.10.015. Epub 2015 Oct 30. PMID 26524704
- [Background] Westfall TC, Westfall DP. Neurotransmission: The Autonomic and Somatic Motor nervous Systems. Pharmacological Basis of Therapeutics, 12th Edition, 171-218, McGraw-HILL, 2011.
- [Background] Standaert DG, Roberson ED. Treatment of Central Nervous System Degenerative Disorders. Pharmacological Basis of Therapeutics, 12th Edition, 609-628, McGraw-HILL, 2011.
- [Background] Lim JH, Wickremasinghe SS, Xie J, Chauhan DS, Baird PN, Robman LD, Hageman G, Guymer RH. Delay to treatment and visual outcomes in patients treated with anti-vascular endothelial growth factor for age-related macular degeneration. Am J Ophthalmol. 2012 Apr;153(4):678-86, 686.e1-2. doi: 10.1016/j.ajo.2011.09.013. Epub 2012 Jan 14. PMID 22245460

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Once Daily | 3 Times Daily
Started | 10 | 10
Completed | 10 | 7
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Once Daily: carbidopa-levodopa 25-100 mg tablets once daily hs for up to 32 days in patients naive to anti-vascular endothelial growth factor (VEGF) injections
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
- 3 Times Daily: carbidopa-levodopa 25-100 mg tablets 3 times daily,in the morning, with supper and hs for up to 32 days in patients naive to anti-VEGF injections
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
- Total: Total of all reporting groups
Arm/Group | Once Daily | 3 Times Daily | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 10 | 5 | 15
Age, Continuous [Mean (Full Range); unit: years] | 76.4 [71 to 81] | 74.1 [58 to 87] | 75.5 [58 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 7 | 17
Patients naive to anti-VEGF injections at start of study [Count of Participants; unit: Participants] | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity
Description: This outcome is a measure of letters correctly identified using an Early Treatment Diabetic Retinopathy Study chart. The higher the number of letters identified, the better the participant's visual acuity.
Time Frame: From start of study to first anti-vascular endothelial growth factor (VEGF) injection (8-32 days)
Population: Statistical comparisons between these two dosages were not completed given the design of this exploratory study. Our publication published findings based on overall exposure to levodopa but did take into account potential adverse effects associated with higher dose frequency of levodopa.
Measure: Mean (Standard Error); unit: Change in letters (BCVA)
Groups:
- Carbidopa/Levodopa Once Daily: carbidopa-levodopa 25-100 mg tablets once daily at bedtime for up to 32 days in patients naive to anti-VEGF injections.
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
- Carbidopa/Levodopa Three Times Daily: carbidopa-levodopa three times daily for up to 32 days in patients naive to anti-VEGF injections.
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
Arm/Group | Carbidopa/Levodopa Once Daily | Carbidopa/Levodopa Three Times Daily
Number analyzed (Participants) | 10 | 7
Change in letters (BCVA) | 6.0 (1.9) | 4.6 (1.6)

2. Secondary Outcome: Change in Central Retinal (Macular) Thickness
Description: Central retinal thickness (in microns) is measured by spectral domain-optical coherence tomography. An increase in retinal thickness is associated with disease progression. A negative value represents a decrease in retinal thickness and therefore a positive clinical outcome measure.
Time Frame: From start of study to first anti-VEGF injection (8-32 days).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microns
Groups:
- Carbidopa/Levodopa Daily: carbidopa-levodopa 25-100 mg tablets once daily for up to 32 days in patients naive to anti-VEGF injections
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
- Carbidopa/Levodopa Three Times Daily: carbidopa-levodopa 25-100 mg tablets three times daily for up to 32 days in patients naive to anti-VEGF injections
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
Arm/Group | Carbidopa/Levodopa Daily | Carbidopa/Levodopa Three Times Daily
Number analyzed (Participants) | 10 | 7
microns | -26.3 (13.4) | -10.3 (10.9)

3. Secondary Outcome: Percent Change in Retinal Fluid From Baseline
Description: Retinal fluid changes on direct retinal examination on spectral domain - optical coherence tomography. Changes in retinal fluid were compared to baseline values. A negative percentage point represents a decrease in retinal fluid and therefore a positive clinical outcome.
Time Frame: From start of study to first anti-VEGF injection (8-32 days)
Measure: Mean (Standard Error); unit: percent change
Groups:
- Carbidopa/Levodopa Daily: carbidopa-levodopa 25-100 mg tablets once daily for up to 32 days on patients naive to anti-VEGF injections.
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
- Carbidopa/Levodopa Three Times Daily: carbidopa-levodopa 25-100 mg tablets three times daily for up to 32 days on patients naive to anti-VEGF injections.
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
Arm/Group | Carbidopa/Levodopa Daily | Carbidopa/Levodopa Three Times Daily
Number analyzed (Participants) | 10 | 7
percent change | -26.4 (11.7) | -32.4 (13.5)

4. Secondary Outcome: Treatment Emergent Adverse Events
Description: Vital signs, eye examinations and nondirected subjective adverse events
Time Frame: From start of study to first anti-VEGF injection (8-32 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Carbidopa/Levodopa Daily: carbidopa-levodopa 25-100 mg tablets once daily hs for up to 32 days in patients naive to anti-VEGF injections
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
Arm/Group | Carbidopa/Levodopa Daily | Carbidopa/Levodopa Three Times Daily
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse event reporting was based on participant-reported systemic adverse events during each study visit. The goal of evaluating differences in once daily and three times daily dosing was to evaluate potential differences in the tolerance/safety of both arms. This is the only secondary outcome that evaluated total daily dose differences of carbidopa/levodopa.
Groups:
- Carbidopa/Levodopa Once Daily: carbidopa-levodopa 25-100 mg tablets once daily hs for up to 32 days in patients naive to anti-VEGF injections.
  carbidopa-levodopa 25-100 mg tablets: See arm/group descriptions
- Carbidopa/Levodopa Three Times Daily: carbidopa-levodopa 25-100 mg tablets three times daily for up to 32 days in patients naive to anti-VEGF injections.
Arm/Group | Carbidopa/Levodopa Once Daily | Carbidopa/Levodopa Three Times Daily
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 1/10 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbidopa/Levodopa Once Daily (N=10) | Carbidopa/Levodopa Three Times Daily (N=7)
Ear issues (Ear and labyrinth disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The major limitations of our study include the small sample size and limited patient racial diversity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-06-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03022318/Prot_001.pdf